CLINICAL TRIAL: NCT02270411
Title: Development of a Method to Isolate Inflammatory Cells From Skin Biopsies of Patients With Various Pathologies for Quantitative Flow Cytometry Analysis
Brief Title: Inflammatory Cells From Various Pathologies
Status: Completed | Type: Observational
Sponsor: Innovaderm Research Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: Inno-6036
Record Dates: First submitted 2014-10-17; First posted 2014-10-21 (Estimated); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Atopic Dermatitis; Acne Rosacea; Acne Vulgaris
MeSH Terms: conditions — Dermatitis, Atopic; Rosacea; Acne Vulgaris

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (6):
- Healthy Subjects: Healthy subjects.
- Atopic Dermatitis: Patient has a history of atopic dermatitis for at least 6 months. Subject has clinically confirmed diagnosis of active atopic dermatitis, according to Hanifin and Rajka criteria.
- Acne Rosacea: Patient has a history of acne rosacea for at least 6 months.
- Acne Vulgaris: Patient has a history of acne vulgaris for at least 6 months.
- Psoriasis: Patient has a history of psoriasis for at least 6 months.
- Hidradenitis Suppurativa (HS): Patient has a history of HS for at least 6 months.

SUMMARY:
The objective of this experiment is to develop and validate in vitro methods to isolate inflammatory cells from skin biopsies for quantitative flow cytometry analysis. Real-time polymerase chain reaction (RT-PCR) will also be performed using skin biopsy samples to validate flow cytometry results. Such methods could eventually be used to better understand the pathophysiology and the mechanism of action of various medications in patients with atopic dermatitis, acne rosacea or vulgaris, HS, and systemic sclerosis.

In this study, up to 15 healthy volunteers, 50 patients with atopic dermatitis, 15 patients with acne rosacea, 15 patients with psoriasis (to be used as control), 15 patients with acne vulgaris, 10 patients with psoriasis to develop a method of analysis for systemic sclerosis, and 10 patients with HS will be recruited.

For the healthy volunteers, atopic dermatitis, psoriasis and HS groups, at least one (1) and a maximum of four (4) skin biopsies (4-5 mm) per subject will be performed. Biopsies will be performed on either the trunk or the limbs, excluding the hands and the feet.

At least one (1) and a maximum of three (3) skin biopsies (2-3 mm) per subject will be collected for the acne rosacea and acne vulgaris groups from one or more body location(s) affected by the pathology.

For patients with atopic dermatitis, an optional blood draw of up to 10 mL will be collected to measure serum IgE levels. For patients with atopic dermatitis, psoriasis, and HS, an optional blood collection of up to 50 mL will be collected to perform flow cytometry on circulating blood cells to study differences in flow cytometry results between cells extracted from biopsies and circulating cells.

DETAILED DESCRIPTION:
Innovaderm, in collaboration with "The Immunoregulation laboratories of CRCHUM" and "McGill University division of dermatology", recently developed a novel 6-hour method to study IL-17A (Interleukin) and IL-22 from fresh biopsies of psoriatic patients. This reproducible experimental approach combines enzymatic digestion and mechanical dissociation for skin cell isolation. This is followed by a multi-color flow cytometry analysis in the absence of in vitro expansion and re-stimulation. Using this method, we examined the cellular source of IL-17A and IL-22 on a small number (20x10³) of viable CD45+ (Cluster of Differentiation Antigen 45) cells that are freshly isolated from 4 mm punch skin biopsies (n=22 patients with psoriasis). The method was used for the study on "Persistence of IL-17A+ T lymphocytes and IL-17A expression in psoriatic plaques refractory to ustekinumab therapy" presented during the 72nd annual meeting of the American Academy of Dermatology in Denver. A detailed presentation of this method will be done during the upcoming annual meeting of the Society for Investigative Dermatology in Albuquerque, New Mexico.

We would like to investigate and adapt this method for other dermatological conditions such as Atopic Dermatitis, Acne Rosacea and Acne Vulgaris.

ELIGIBILITY:
Inclusion Criteria:

* Subject, male or female, is aged 18 years or older at the screening visit.
* Female subjects of childbearing potential must have a negative urine pregnancy test at the Screening visit.
* Subjects must be able and willing to provide written informed consent and comply with the requirements of this study protocol.

  **Special inclusion criterion for volunteers with atopic dermatitis, acne rosacea, acne vulgaris, psoriasis, or HS
* Patient has a history of atopic dermatitis, acne rosacea, acne vulgaris, psoriasis, or HS for at least 6 months.

  **Special inclusion criterion for volunteers with atopic dermatitis
* Subject has clinically confirmed diagnosis of active atopic dermatitis, according to Hanifin and Rajka criteria

Exclusion Criteria:

* Female subject is pregnant or lactating
* Subject is currently participating in a clinical trial with an experimental drug or device
* Subject is known to have hepatitis B or hepatitis C viral infection
* Subject is known to have immune deficiency or is immunocompromised
* Subject has a known hypersensitivity/allergy to lidocaine
* Patient has a history of keloids
* Patient is taking heparin, warfarin or has a contraindication to skin biopsies.
* Patient has used systemic medication, medical devices or natural health products to treat acne rosacea, atopic dermatitis, acne vulgaris, psoriasis, or HS, or UVB phototherapy within 4 weeks of biopsy day
* Patient has used oral, intravenous, intramuscular or intra-lesional or intra-articular steroids, or immunosuppressive medication within 4 weeks of biopsy day
* Patient has used a biologic agent within 24 weeks or 5 half-lives (whichever is longer) of biopsy day
* Patient has used topical medication, natural health products or medical devices to treat acne rosacea, atopic dermatitis, acne vulgaris, psoriasis, or HS on the areas to be biopsied within 2 weeks of biopsy day
* Patients is currently using or has used isotretinoin

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Invitation to volunteer
Sampling Method: Non-Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2014-05; Primary Completion 2023-12 (Actual); Study Completion 2023-12 (Actual)

PRIMARY OUTCOMES:
Proportion of Inflammatory Cells in Skin Biopsies | 1 Day
  The proportion of inflammatory cells in skin biopsies will be assessed by flow cytometry.

SECONDARY OUTCOMES:
Expression of Inflammation-Related Genes in Skin Biopsies | 1 Day
  The level of expression of inflammation-related genes in skin biopsies will be assessed by quantitative real-time polymerase chain reaction (qRT-PCR).

CONTACTS AND LOCATIONS:
Overall Officials: Robert Bissonnette, MD, Principal Investigator — Innovaderm Research
Locations (1):
- Innovaderm Research, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No